CLINICAL TRIAL: NCT02218762
Title: A Randomised, Two Treatment, Four-Way Cross-Over (Replicate Design), Two Sequence, Repeat Dose Study in Patients With Moderate Asthma to Compare Pharmacokinetics and Pharmacodynamic Effects of Fluticasone Propionate and Salmeterol Delivered Via the Low Airflow Resistance Fluticasone Propionate/Salmeterol (100/50 mcg) ROTAHALER Inhaler Relative to Fluticasone Propionate/Salmeterol (100/50 mcg) Delivered Via the DISKUS Inhaler
Brief Title: A Study in Patients With Moderate Asthma to Compare Pharmacokinetics and Pharmacodynamic Effects of Fluticasone Propionate and Salmeterol Delivered Via the ROTAHALER® Inhaler Relative to the DISKUS® Inhaler
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: It was decided that data from this study are no longer required and therefore it is not necessary to expose patients to the study medication
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201461
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Asthma
Keywords: Fluticasone propionate/salmeterol in a capsule-based inhaler; replicated cross-over design; Respiratory; asthma; safety; pharmacokinetics; Fluticasone propionate/salmeterol; pharmacodynamics; Fluticasone propionate/salmeterol in a multi-dose dry powder inhaler
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects will receive FSC 100/50 mcg delivered via the Ddpi (Treatment A) and FSC 100/50 mcg delivered via the Rdpi (Treatment B) in the sequence of A-B-B-A in four treatment periods of 10 days each. Subjects will receive both active treatment and matching placebo at the same time from two separate devices twice daily. There will be no wash-out between treatment periods
  Interventions: Drug: Fluticasone Propionate/Salmeterol Xinafoate DISKUS; Drug: Placebo to Match DISKUS; Drug: Fluticasone Propionate/Salmeterol Xinafoate ROTACAPS; Drug: Placebo to Match ROTACAPS
- Sequence 2 (Experimental): Subjects will receive FSC 100/50 mcg delivered via the Ddpi (Treatment A) and FSC 100/50 mcg delivered via the Rdpi (Treatment B) in the sequence of B-A-A-B in four treatment periods of 10 days each. Subjects will receive both active treatment and matching placebo at the same time from two separate devices twice daily. There will be no wash-out between treatment periods
  Interventions: Drug: Fluticasone Propionate/Salmeterol Xinafoate DISKUS; Drug: Placebo to Match DISKUS; Drug: Fluticasone Propionate/Salmeterol Xinafoate ROTACAPS; Drug: Placebo to Match ROTACAPS

INTERVENTIONS:
Drug: Fluticasone Propionate/Salmeterol Xinafoate DISKUS — A blister strip contained within the DISKUS inhaler. Each blister contains a small quantity of powder comprising of a blend of fluticasone propionate (micronized)(100 mcg), salmeterol xinafoate (micronized) (50 mcg) and excipient(s). One blister to be administered twice daily via DISKUS inhaler
Drug: Placebo to Match DISKUS — A blister strip contained within the DISKUS inhaler. Each blister contains a small quantity of lactose and powder comprising of excipient(s). One blister to be administered twice daily via DISKUS inhaler
Drug: Fluticasone Propionate/Salmeterol Xinafoate ROTACAPS — A capsule containing a small quantity of powder comprising of a blend of fluticasone propionate (micronized) (100 mcg), salmeterol xinafoate (micronized) (50 mcg) and excipient(s). One capsule to be administered twice daily via ROTAHALER inhaler
Drug: Placebo to Match ROTACAPS — A capsule containing a small quantity of lactose and powder comprising of excipient(s). One capsule to be administered twice daily via ROTAHALER inhaler

SUMMARY:
The Fluticasone Propionate/Salmeterol combination (FSC) at a dose of 100/50 micrograms (mcg) twice daily in DISKUS inhaler (also known as ACCUHALER®, Ddpi) inhaler is a recognised and licensed therapy for the treatment of asthma. GlaxoSmithKline (GSK) is developing the ROTAHALER/ ROTACAPS® (Rdpi) inhaler as an alternative treatment option for asthmatic patients. This study is a Phase I, randomised, double-blind, double-dummy, two- treatment, four-way cross-over (replicate design), two sequence, repeat dose, two centre study in mild to moderate asthmatics to compare the pharmacokinetics and pharmacodynamics of fluticasone proprionate/salmeterol (100/50 mcg) delivered via the Rdpi versus the Ddpi. A total of 58 subjects will be enrolled to ensure 52 subjects complete all dosing occasions. Each subject will be allocated to one of two treatment sequences and will participate in four treatment periods, receiving each of the treatments twice.

DISKUS, ACCUHALER, ROTAHALER and ROTACAPS are registered trademarks of GSK groups of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a known physician diagnosis of asthma with a best Forced Expiratory Volume in 1 Second (FEV1) of >70% of the predicted normal value at the Screening visit. Percent predicted will be calculated using the European Respiratory Society Global Lung Function Initiative reference equations. Subjects must abstain from short acting beta-2 agonists (SABA) use for 6 hours prior to the Screening visit.
* During the screening visit, subjects must either demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of >=12.0% over baseline and an absolute change of >=200 millilitres (mL) within 60 minutes following 4 inhalations of albuterol/salbutamol inhalation aerosol (or equivalent nebulized treatment with albuterol/salbutamol solution) or in the absence of reversibility have documented evidence of a physician diagnosed asthma for at least 6 months
* Male/females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight >= 50 kilograms (kg) and body mass index (BMI) within the range 18 - 35.0 kilogram/square meter (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milliinternational units per/millilitre (MIU/mL) and estradiol <40 picogram/millilitre (pg/mL) (<147 picomoles per liter [pmol/L]) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.; Child-bearing potential with negative pregnancy test as determined by serum or human chorionic gonadotropin (hCG) test at screening or urine hCG test prior to dosing AND ; Agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.; OR has only same-sex partners, when this is her preferred and usual lifestyle.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Subjects who are current non-smokers and who have a pack history of <=10 pack years. A subject may not have used inhaled tobacco products within the past 3 months (i.e., cigarettes, cigars or pipe tobacco). [number of pack years = (number of cigarettes per day / 20) x number of years smoked].
* Alanine transaminase (ALT), alkaline phosphatase and bilirubin <= 1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiogram (ECGs) obtained over a brief recording period: QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (msec); or QTcF <480 msec in subjects with Bundle Branch Block.
* Asthma therapy: Subjects must have been on their current therapy for at least eight weeks and a stable dose for four weeks prior to the screening visit:

  1. Subjects on fluticasone propionate/salmeterol combination 100/50 microgram (mcg) treatment via a DISKUS inhaler prior to the study will be allowed to remain on their treatment regimen until randomization provided all other eligibility criteria are met.;
  2. Subjects on treatment with fluticasone propionate/salmeterol combination 125/25 mcg via a metered dose inhaler will be required to switch to fluticasone propionate/salmeterol combination 100/50 mcg via the GlaxoSmithkline (GSK)-provided DISKUS inhaler for between 14 and 28 days prior to randomization;
  3. Subjects on low dose inhaled corticosteriod (ICS) monotherapy (up to a total daily dose of fluticasone propionate 250 total daily dose mcg or other ICS equivalent e.g. budesonide up to 400 mcg total daily dose) will switch to fluticasone propionate/salmeterol combination 100/50 mcg via the GSK-provided DISKUS inhaler for between 14 and 28 days prior to randomization;
  4. Subjects on medium dose ICS monotherapy ( greater than 250 and up to 500 mcg of fluticasone propionate total daily dose or other ICS equivalent e.g. budesonide greater than 400 mcg and up to 800 mcg total daily dose) will switch to fluticasone propionate/salmeterol combination 100/50 mcg twice daily via the GSK-provided DISKUS inhaler for 28 days prior to randomization;
  5. Subjects on low dose Symbicort (any doses that are no greater than 400/12 mcg total daily dose) will be switched to fluticasone propionate/salmeterol combination 100/50 mcg via the GSK-provided DISKUS inhaler for between 14 and 28 days prior to randomization.

Exclusion Criteria:

Criteria Based Upon Medical Histories

* Any clinically relevant medical condition or abnormality identified during the screening medical assessment and procedures, physical examination, or laboratory assessments (including clinical chemistry and haematology), which in the opinion of the Investigator and/or GSK Medical Monitor is likely to affect the safety of the subject and/or interfere with the study procedures and outcomes.
* Acute exacerbation of asthma in the last 6 months prior to the Screening visit.
* Subjects on treatment with fluticasone propionate either as monotherapy or in combination at a total daily dose higher than 500 mcg or budesonide monotherapy or in combination at a total daily dose higher than 800 mcg or beclomethasone (CFC) at a total daily dose higher than 1000 mcg or beclomethasone (HFA) at a total daily dose higher than 400mcg are excluded from the study
* Subjects with other significant pulmonary diseases (pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma).
* Use of oral/injectable/depot corticosteroid for any indication within 3 months prior to the Screening visit.
* Use of any anti immunoglobulin E (Anti-IgE) (e.g. Xolair) in any period prior to screening.
* Use of intra-nasal steroids (INS). To be eligible for the study, patients on INS therapy will be required to switch to non-INS therapy at screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: For Australian sites: An average weekly intake of >21 units for males or >14 units for females. One unit (= standard drink) is equivalent to 10 g of alcohol: 270 mL of full strength beer (4.8%), 375 mL of mid strength beer (3.5%), 470 mL of light beer (2.7%), 250 mL pre-mix full strength spirit (5%), 100 mL of wine (13.5%) and 30 mL of spirit (40%); For South African sites: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 330 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* A known or suspected history of drug abuse within 12 months of the Screening visit.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to salbutamol or any of the study medications, or components thereof (including severe milk protein allergy) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Subjects with known abnormal levels of serum cortisol
* A subject will not be eligible if he/she has clinical visual evidence of oral candidiasis prior to randomisation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Grapefruit or grapefruit juice containing products are excluded from 2 weeks prior to randomisation until collection of the final blood sample at treatment period 4.
* Drugs that inhibit the cytochrome P450 isoform, 3A4 (CYP3A4), are excluded from 2 weeks prior to randomisation until collection of the final blood sample at treatment period 4. CYP3A4 inhibitors include cimetidine, clarithromycin, erythromycin, ciprofloxacin, ritonavir, ketoconazole, and azole antifungals.
* Use of prescription or non-prescription drugs, vitamins, herbal and dietary supplements, within seven days or 5 half-lives (whichever is longer) prior to the first dose of study medication, which in the opinion of the Principal Investigator, may interfere with study outcome. Specifically, calcium and vitamin D supplements and bisphosphonates are not allowed throughout the study.
* Subjects, who, in the opinion of the Investigator, are not able to comply with the protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Fluticasone propionate (FP) area under the concentration-time curve over the dosing interval (AUCtau) | Day 10 of each treatment period (pre-morning dose and at 5, 10, 30 minutes and 1, 2, 4, 8, 10 and 12 hours post- morning dose)
  FP AUCtau will be determined from the plasma FP concentration-time data
Salmeterol maximum observed concentration (Cmax) | Day 10 of each treatment period (pre-morning dose and at 5, 10, 30 minutes and 1, 2, 4, 8, 10 and 12 hours post- morning dose)
  Salmeterol Cmax will be determined from the plasma salmeterol concentration-time data

SECONDARY OUTCOMES:
Salmeterol AUCtau | Day 10 of each treatment period (pre-morning dose and at 5, 10, 30 minutes and 1, 2, 4, 8, 10 and 12 hours post- morning dose)
  Salmeterol AUCtau will be determined from the plasma FP concentration-time data
FP Cmax | Day 10 of each treatment period (pre-morning dose and at 5, 10, 30 minutes and 1, 2, 4, 8, 10 and 12 hours post- morning dose)
  FP Cmax will be determined from the plasma FP concentration-time data
FP and salmeterol time to Cmax (Tmax) | Day 10 of each treatment period (pre-morning dose and at 5, 10, 30 minutes and 1, 2, 4, 8, 10 and 12 hours post- morning dose)
  FP and salmeterol Tmax will be determined from the plasma FP concentration-time data
Weighted mean serum cortisol over 12 hours on the last day of each treatment period (Day 10) | Day 10 of each treatment period
  Blood sampling for measurement of serum cortisol will be performed on the last day of each treatment period (Day 10) at pre-morning dose and at 30 min, 1,2,4,8,10 and 12 hours post- morning dose. Weighted mean concentration from 0 to 12 hours will be derived from the serum cortisol concentration data
Serum cortisol minimum observed concentration (Cmin) | Day 10 of each treatment period
  Blood sampling for measurement of serum cortisol will be performed on the last day of each treatment period (Day 10) at pre-morning dose and at 30 min, 1,2,4,8,10 and 12 hours post- morning dose. Cmin will be derived from the serum cortisol concentration data
Heart rate (HR) measurements | Up to 10 weeks
Blood pressure (BP) measurements | Up to 10 weeks
  Systolic and diastolic blood pressure will be measured
Potassium and Glucose measurements | Up to 10 weeks
  Blood sampling for measurement of potassium and glucose will be performed on Day 1 Treatment Period 1 (pre-dose) and on Day 10 of each treatment period (pre-morning dose and at 30, 60 minutes, 2 and 4 hours post the morning dose)
Number of subjects with adverse events | Up to 12 weeks
  An adverse event is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Clinical laboratory safety assessments | Up to 12 weeks
  Haematology, clinical chemistry, and urinalysis parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline